CLINICAL TRIAL: NCT00795028
Title: Preventing Falls and Disability in Older Adults After Hip Fracture
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Maureen C. Ashe, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: H08-01685
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Hip Fracture
Keywords: older women; hip fracture; exercise intervention
MeSH Terms: conditions — Hip Fractures | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard Care for people after a hip fracture
  Interventions: Other: Standard Care for people after hip fracture
- 2 (Experimental): Standard Care + exercise intervention
  Interventions: Other: Standard Care + exercise intervention

INTERVENTIONS:
Other: Standard Care for people after hip fracture
  Arms: 1
Other: Standard Care + exercise intervention
  Arms: 2

SUMMARY:
Patients who have suffered a first hip fracture have a higher risk of falling and sustaining another hip fracture compared with age-matched adults who did not fracture. Although exercise is key to reversing this pattern, there have been very few trials that aimed to improve muscle strength and balance as well as enhance bone health following hip fracture. Therefore, we propose to conduct an RCT that delivers either 12 months of standard care or standard care plus graduated exercise program for older women who have sustained a recent hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* Older community dwelling women who have sustained a first hip fracture

Ages: 65 Years to 105 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Fall rate, measured by self-reported daily fall diaries, will be collected monthly at the exercise classes and followed up by an independent investigator | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: M C Ashe, PhD, Principal Investigator — University of British Columbia